CLINICAL TRIAL: NCT05402072
Title: Autologous MatRix-Induced ChondrogenEsis ComPared With Microfracture for Focal ArtIcular CaRtilage Damage of the Hip (REPAIR): A Pilot Randomized Controlled Trial
Brief Title: AMIC Compared With Microfracture for Focal Articular Cartilage Damage of the Hip
Acronym: REPAIR
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Geistlich Pharma AG (Industry)
Responsible Party: Principal Investigator, Olufemi Ayeni, Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 14981
Record Dates: First submitted 2022-05-25; First posted 2022-06-02 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Hip Arthroscopy; Articular Cartilage Defect; Microfractures
MeSH Terms: conditions — Fractures, Stress

STUDY DESIGN:
Intervention Model Description: All patients presenting to each clinical site's out-patient fracture clinics and/or sports medicine subspecialty clinics between ages of 18 and 5 years with a symptomatic chondral injury of the hip will be screened. There will be a Research Coordinator on hand during the initial phase of the surgery for each consented patient, where the surgeon will assess the final aspects of eligibility. If eligibility is confirmed, the Research Coordinator will randomize the patient using a centralized 24-hour online randomization system that will follow a randomization schedule in random block sizes of 4 and 8. The secure online randomization system will ensure concealment of the treatment allocation. If the surgeon deems intra-operatively that the subject does not meet the inclusion criteria, the surgeon will manage the lesion as per the normal standard of care and the subject's ineligibility will be recorded on the screening form.
Who Masked: Participant, Outcomes Assessor
Masking Description: The outcome assessors, those performing data entry and analysis, and patients will be blinded to the treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Microfracture (Active Comparator): As per current standard of care for focal articular cartilage lesions of the acetabulum, the unstable cartilage will be debrided and removed from the subchondral bone using a mechanical shaver until a stable margin is obtained. A ring curette will be used to remove the calcified cartilage layer and create a border of healthy cartilage tissue that can support the marrow clot. Through the mid-anterior portal, specialized 90˚ awls will then be placed with the tip perpendicular to the subchondral bone of the acetabulum, and a mallet will be used to penetrate the subchondral bone with perforations 3 mm deep to access the bone marrow elements. This is done until the defect is homogeneously covered with micro-perforations 2-3 mm apart.
  Interventions: Procedure: Autologous matrix-induced chondrogenesis (AMIC)
- Autologous matrix-induced chondrogenesis (AMIC) (Experimental): Those allocated to the AMIC treatment group will also receive microfracture. Once the walls of the debrided lesion are confirmed to be stable with a probe, the exact size of the defect will be measured for templating of the scaffold. The dry Chondro-Gide® matrix will be prepared by cutting it to 10% smaller than the focal defect (as it increases in size about 10% after moistening). Once the cartilage lesion is dried manually, the implant will then be secured to the defect in a press-fit fashion to the surrounding cartilage. Manual pressure is then applied to secure the implant into the defect and the hip is released from traction and rotated to facilitate further fixation of the graft. Traction is then applied to arthroscopically confirm position and fixation of the implant.
  Interventions: Procedure: Autologous matrix-induced chondrogenesis (AMIC)

INTERVENTIONS:
Procedure: Autologous matrix-induced chondrogenesis (AMIC) — AMIC is a novel approach in which the microfracture technique has been enhanced by the use of a type I/III collagen matrix (Chondro-Gide®; Geistlich Pharma AG, Wolhusen, Switzerland). In this single-step procedure, the matrix is placed over the defect to stabilize the fragile blood clot that arises from microfracture and to provide infrastructure for repair tissue formation. Essentially, the matrix covers the defect and serves as a protective shield that contains the cells and minimizes the impact of shear forces when moving the hip on the delicate blood clot. At the same time, it functions as the roof of a biological chamber that forms over the defect. The biocompatible collagen material provides an environment for cell growth and is replaced by native tissue over time.
  Other Names: Chondro-Gide(R)

SUMMARY:
This is a pilot multi-centre RCT of 40 patients (ages 18-55 years, inclusive) undergoing primary hip arthroscopy with a focal articular cartilage defect of the acetabulum to compare the effect of using autologous matrix-induced chondrogenesis (AMIC) in comparison to microfracture on hip function, health-related quality of life, hip pain, cartilage regeneration, health utility, and any adverse events at 2 years. Follow-up will occur at 6 weeks, 6 months, 12 months, 18 months, and 24 months post-surgery.

ELIGIBILITY:
Inclusion Criteria:

1. All patients aged 18-55 years
2. Hip pain lasting 6 months or more with no relief from documented non-operative modalities
3. Focal articular cartilage defects of the acetabulum on MRI, confirmed to be full thickness (International Cartilage Regeneration and Joint Preservation Society (ICRS) grade 3 or 4) during arthroscopic examination
4. Focal acetabular articular cartilage lesions measuring between 3 cm2 and 25 cm2 on MRI and confirmed on arthroscopic examination
5. Patient agrees to participate in the study-specific postoperative rehabilitation protocol
6. Patient can speak, read, and understand the language of the site
7. Patient has provided informed consent

Exclusion Criteria:

1. Cartilage defects of the femoral head
2. Previous surgery on the study hip
3. Traumatic chondral injury of the hip from a single event
4. Presence of advanced osteoarthritis (Tonnis grade 3) or any other acute or chronic inflammatory joint disease
5. Known hypersensitivity or allergy to porcine collagen
6. Acute or chronic infection at the surgical site
7. Evidence of hip dysplasia (i.e., lateral centre edge angle < 20˚)
8. Evidence of acetabular over coverage such as coxa profunda or coxa protrusion
9. Immunosuppressive or anti-proliferative medication use
10. Chronic pain syndromes
11. Significant medical co-morbidities (requiring assistance for activities of daily living (ADLs))
12. History of paediatric hip disease
13. Uncontrolled diabetes
14. Contraindications to MRI imaging (e.g. claustrophobia)
15. Patient is involved in ongoing legal or workplace claims
16. Patient is incarcerated
17. Patient is pregnant or breastfeeding
18. Patient who will likely have problems, in the judgement of the investigator, with maintaining follow-up
19. Any other reason(s) the investigator feels is relevant for excluding the patient

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-03-13 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Hip function and health-related quality of life using the International Hip Outcome Tool (iHOT-33) | Change from baseline to 24 months post-surgery
  The iHOT-33 is designed to measure hip-specific health-related quality of life changes after treatment of active young patients with hip disorders. The total score is calculated as a simple mean of the responses ranging from 0 to 100, with 100 representing the best possible quality-of-life score.

SECONDARY OUTCOMES:
Hip pain using the Visual Analogue Scale (VAS); 100-point scale | Change from baseline to 24 months post-surgery
  To measure hip pain. The total score is calculated as a single response ranging from 0 to 100, with 100 representing the worst possible pain.
Cartilage repair using the Magnetic Resonance Evaluation of the Repair of Cartilage in the Hip Score (MERCH) (scored from 0-100) | Change from baseline to 24 months post-surgery
  To evaluate cartilage repair in the hip using MRI imaging. The total score is calculated as a simple mean of the responses ranging from 0 to 100, with 0 representing the worst cartilage status.
Health utility using the Euro-Qol 5 Dimensions (EQ-5D); index score | Change from baseline to 24 months post-surgery
  Utility-based instrument for use as a measure of health outcome. Health state index scores generally range from less than 0 (where 0 is the value of a health state equivalent to dead; negative values representing values as worse than dead) to 1 (the value of full health), with higher scores indicating higher health utility.
Total number of adverse events | 24 months post-surgery
  Any reported complications such as infection, additional or revision surgery, hypersensitivity or allergic reactions, and reduced range of motion

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No